CLINICAL TRIAL: NCT06975865
Title: A 52-week, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Group Sequential Study to Evaluate the Efficacy and Safety of Rilzabrutinib in Patients Aged 10 to 65 Years With Sickle-cell Disease
Brief Title: The Efficacy and Safety of Rilzabrutinib in Patients Aged 10 to 65 Years With Sickle-cell Disease
Acronym: LIBRA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17872; 2024-518645-17 (Registry Identifier: CTIS); U1111-1311-1896 (Other Grant/Funding Number: ICTRP)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rilzabrutinib (Experimental): Rilzabrutinib
  Interventions: Drug: Rilzabrutinib
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilzabrutinib — Pharmaceutical form:Tablet -Route of administration:Oral
  Other Names: SAR444671
  Arms: Rilzabrutinib
Drug: Placebo — Pharmaceutical form:Tablet -Route of administration:Oral
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, group-sequential study (Part A), followed by an open-label LTE period (Part B) to investigate the efficacy, and safety of rilzabrutinib in participants with sickle-cell disease (SCD).

Study details include:

* Study duration: a 52-week double-blind period (Part A), followed by an open-label LTE period (Part B). Double-blind period has two parts, 50% (adult only) until the interim analysis (a proof-concept part analogous to a phase 2b study), and 50% (adult and children) after the interim analysis. Only the participants who complete double-blind treatment period (Part A) are eligible to continue to the LTE period. The duration of the LTE period (Part B) will be from the first-participant-in (FPI)-LTE (Part B) until the last participant who enters the LTE has completed 52 weeks.
* Treatment duration: 52-week double-blind period (Part A); LTE period (Part B) from the (FPI until the last participant who enters the LTE has completed 52 weeks.
* Visit frequency: Week visits based on the Schedule of Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been diagnosed with SCD.
* Participants who have had between ≥2 to ≤10 episodes of documented acute clinical VOC within 12 months of the screening visit.
* Participants who are either not on hydroxyurea and/or L-glutamine at the Screening Visit and does not plan to receive them during the course of the study or has received HU and/or L-glutamine for a minimum of 6 months. Participants on hydroxyurea and/or L-glutamine must have been on a stable weight-based dose level (mg/kg) for at least 3 months prior to the Screening Visit, with the intent to continue at the same weight-based dose level for the duration of the study, except for safety reasons.
* Participants with Eastern Cooperative Oncology Group (ECOG) performance status grade 2 or lower.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* For participants ≥10 to <18 years of age: the parent(s)/legal guardian(s) must provide written informed consent prior to any study-related procedures being performed.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply: Participants with medical history of lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for the past 3 years.
* Clinically relevant cardiac abnormality, in the opinion of the Investigator or electrocardiogram (ECG) findings.
* Participants with history of stroke, or history of abnormal transcranial doppler.
* Participants with uncontrolled or active HBV infection and/or HCV infection including those receiving antiviral therapy at the time of screening.
* HIV infection.
* A history of active or latent tuberculosis (TB)
* Positive COVID-19 molecular test.
* Participant is taking or has received crizanlizumab (ADAKVEO®) within 90 days and/or voxelotor (OXBRYTA®) within 30 days prior to the Screening visit.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-07-23 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of clinical VOC | At Week 52
  Calculated from total number of clinical VOC incidents and total number of days during the observation period

SECONDARY OUTCOMES:
Time to first clinical VOC incidence | Until Week 52
Annualized rate of visits due to SCD-related complications as assessed by the Investigator | At Week 52
Annualized rate of home-managed VOCs as reported in the Sickle Cell Pain Crisis (SCPC) eDiary | At Week 52
Change in fatigue as measured by the PROMIS SF v1.0 Fatigue 13a total score (adults) | From baseline to Week 52
Change in Hb levels | From baseline to Week 52
Change in fatigue as measured by the PedsQL Multidimensional Fatigue Scale total score (pediatric participants) | From baseline to Week 52
Incidence of treatment emergent adverse events (TEAEs), including serious adverse events (SAEs), adverse events of special interest (AESIs) and adverse events leading to discontinuation | Until Week 52
Incidence of potentially clinically significant laboratory, vital signs, and ECG abnormalities | Until Week 52
Absolute number of simple and exchange blood transfusion | Until Week 52
Number of days requiring acetaminophen, NSAID and/or short-acting opioid usage | Until Week 52

CONTACTS AND LOCATIONS:
Locations (46):
- United States (8):
  - University of Alabama at Birmingham- Site Number : 8400003, Birmingham, Alabama
  - Oncology & Hematology Associates of West Broward- Site Number : 8400029, Coral Springs, Florida
  - Louisiana State University Health Sciences Center - Shreveport- Site Number : 8400037, Shreveport, Louisiana
  - University of Michigan Health System - Ann Arbor- Site Number : 8400035, Ann Arbor, Michigan
  - Southern Specialty Research- Site Number : 8400059, Flowood, Mississippi
  - Richmond University Medical Center- Site Number : 8400038, Staten Island, New York
  - Baylor College of Medicine- Site Number : 8400055, Houston, Texas
  - VCU Massey Cancer Center: Dalton Oncology Clinic- Site Number : 8400012, Richmond, Virginia
- Belgium (3):
  - Investigational Site Number : 0560003, Brussels
  - Investigational Site Number : 0560002, Brussels
  - Investigational Site Number : 0560001, Leuven
- Brazil (5):
  - Hospital Santa Izabel- Site Number : 0760006, Salvador, Estado de Bahia
  - Universidade Federal da Bahia - Site Number : 0760009, Salvador, Estado de Bahia
  - Universidade Federal de Goias- Site Number : 0760002, Goiânia, Goiás
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto- Site Number : 0760001, São José do Rio Preto, São Paulo
  - Hospital Samaritano De Sao Paulo- Site Number : 0760005, São Paulo
- France (4):
  - Investigational Site Number : 2500002, Créteil
  - Investigational Site Number : 2500005, Marseille
  - Investigational Site Number : 2500001, Paris
  - Investigational Site Number : 2500004, Toulouse
- Ghana (2):
  - Investigational Site Number : 2880004, Kintampo
  - Investigational Site Number : 2880002, Navrongo
- Greece (3):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000003, Athens
  - Investigational Site Number : 3000002, Pátrai
- Israel (4):
  - Investigational Site Number : 3760001, Afula
  - Investigational Site Number : 3760002, Afula
  - Investigational Site Number : 3760005, Haifa
  - Investigational Site Number : 3760006, Haifa
- Italy (7):
  - Azienda Ospedaliero Universitaria Careggi SOD Ematologia-Site Number : 3800006, Florence, Firenze
  - Investigational Site Number : 3800004, Milan, Milano
  - Azienda Ospedaliera Universitaria, Università della Campania "Luigi Vanvitelli" Napoli-Site Number : 3800005, Naples, Napoli
  - IRCCS Ospedale Pediatrico Bambino Gesù-Site Number : 3800001, Rome, Roma
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, SSD Microcitemie Malattie Rare Ematologiche-Site Number : 3800007, Orbassano, Torino
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello-Site Number : 3800002, Palermo
  - Centro Ricerche Cliniche Verona s.r.l. presso Ospedale G.B. Rossi Borgo Roma-Site Number : 3800003, Verona
- Investigational Site Number : 5280002, Rotterdam, Netherlands
- Investigational Site Number : 5120001, Muscat, Oman
- Spain (2):
  - Investigational Site Number : 7240002, Madrid
  - Investigational Site Number : 7240001, Madrid
- Investigational Site Number : 8340003, Mwanza, Tanzania
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920001, Adana
  - Investigational Site Number : 7920002, Adana
  - Investigational Site Number : 7920003, Mersin
- United Kingdom (2):
  - Investigational Site Number : 8260002, London, Harrow
  - Investigational Site Number : 8260001, London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17872 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26677&tenant=MT_SNY_9011